CLINICAL TRIAL: NCT05268822
Title: Movement Control Exercises With and Without Specific Breathing Techniques for the Treatment of Chronic Low Back Pain: an Open-label Feasibility Study With 2-month
Brief Title: Movement Control Exercises With and Without Specific Breathing Techniques for the Treatment of Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Jani Mikkonen, Principal Investigator / PhD student at Institute of Clinical Medicine, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KuopioUH_2022
Record Dates: First submitted 2022-02-08; First posted 2022-03-07 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Intervention Model Description: An open-label feasibility study with study subject allocated to movement control exercise with specific breathing techniques (experimental group) or movement control exercise without specific breathing techniques (control group)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement control exercise with specific breathing techniques (Active Comparator): Movement control exercise with specific breathing techniques (experimental group)
  Interventions: Other: Home exercise
- Movement control exercise without specific breathing techniques (Active Comparator): Movement control exercise without specific breathing techniques (control group)
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Home exercise — Movement control exercise with or without specific breathing techniques

SUMMARY:
Chronic low back pain (CLBP) is a leading disability globally. Exercise therapies are one of the most commonly prescribed treatment options for CLBP. Specific breathing techniques have been shown to enhance brain-based pain modulation and autonomic nervous system balance; these changes have been shown to improve clinical effectiveness in terms of pain management and psychological factors compared to general exercise. However, no previous studies have added a specific breathing technique protocol to an evidence-based exercise program for CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-68-years-old
* Low back pain lasting more than 3 months (pain sensation more than 3 days per week)
* A numerical pain scale of more than 3
* ≥ 2/6 positive low back movement control tests (as described by Luomajoki et al.)
* Roland-Morris Disability Questionnaire score of five or greater
* Who are physically able to perform movement control tests and provide written informed consent.

Exclusion Criteria:

* Any history of malignant cancer
* Neurological disease affecting the central nervous system (MS, dementia)
* Rheumatic disease (fibromyalgia, ankylosing spondylitis/rheumatoid arthritis)
* Chronic obstructive pulmonary disease,
* Spinal surgery in the last 12 months
* A cardiac pacemaker
* Signs and symptoms of nerve root pathology during the clinic visits.
* Women who become pregnant during the data collection will also be excluded from the study.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
The numerical pain rating scale (NRPS) | Change from Baseline The numerical pain rating scale at 2 months
  Eleven-point numerical pain scale. Scale from 0 (no pain) to 10 (worst imaginable)
Well-Being in Pain Questionnaire | Change from Baseline Well-Being in Pain Questionnaire at 2 months
  Self-developed questionnaire to screen the effects of pain on a person's biopsychosocial well-being. Scale from 0 (no subjective well-being in pain) to 60 (maximum subjective well-being in pain)
The Roland Morris Disability Questionnaire (RMDQ) | Change from Baseline The Roland Morris Disability Questionnaire at 2 months
  Questionnaire measuring disability in chronic low back pain populations. Scale from 0 (no disability) to 24 (maximum low back pain related disability)
Central Sensitization Inventory (CSI) | Change from Baseline Central Sensitization Inventory at two months
  Screening of central sensitization phenomenon. Scale from 0 (no central sensitization) to 100 (worst imaginable central sensitization)
The 5-level EQ-5D version of the EuroQol | Change from Baseline The 5-level EQ-5D version of the EuroQol at 2 months
  Health status. Scale from 0 (dead) to 1 (full health)
The Generalised Anxiety Disorder Assessment (GAD-7) | Change from Baseline The Generalised Anxiety Disorder Assessment at two months
  Measure of generalised anxiety disorder related symptoms. Scale from 0 (the most minimal anxiety) to 21 (the most severe anxiety)
The Tampa Scale of Kinesiophobia (TSK) | Change from Baseline The Tampa scale of Kinesiophobia at two months
  Assessment of subjective kinesiophobia (fear of movement). Scale from 17 (the minimal kinesophobia) to 68 (the most maximum kinesiophobia).
The Pain Catastrophizing Scale (PCS) | Change from Baseline he Pain Catastrophizing Scale at two months
  Assessment of catastrophizing (tendency to magnify the threat value of a pain stimulus) related to pain. Scale from 0 (no catastrophizing thoughts) to 52 (maximum catastrophizing thoughts)
The Pain and Sleep Questionnaire Three-Item Index (PSQ-3) | Change from Baseline The Pain and Sleep Questionnaire Three-Item Index at two months
  Effect of pain on sleep. Scale from 0 (pain have no any effect on sleep) to 30 (pain have maximum effect on sleep)
The Pain Self-Efficacy Questionnaire (PSEQ) | Change from Baseline The Pain and Sleep Questionnaire Three-Item Index at two months
  assess the self-efficacy of people in pain have in daily activities. The scale is from 0 points (not at all confident) to 6 points (completely confident).

SECONDARY OUTCOMES:
Feasibility of intervention protocol, recruitment and enrollment | Through study completion, an average of 2 mothns
  To assess the feasibility of the intervention protocol and subject recruitment and enrollment.
Responsiveness | Through study completion, an average of 2 months
  To quantify the changes in and determine the responsiveness of the outcome measures, in order to calculate the sample size for a randomized controlled trial (RCT) based on the chosen primary outcome measure(s).
Quantifying | Through study completion, an average of 2 months
  To quantify the changes in self-adherence levels to home exercise and monitor possible pain medication usage, and side effects, adverse events and injuries during exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Private Clinic of principal investigator, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mikkonen J, Luomajoki H, Airaksinen O, Goubert L, Pratscher S, Leinonen V. Identical movement control exercises with and without synchronized breathing for chronic non-specific low back pain:A randomized pilot trial. J Back Musculoskelet Rehabil. 2024;37(6):1561-1571. doi: 10.3233/BMR-230413. PMID 39031339
- [Derived] Mikkonen J, Luomajoki H, Airaksinen O, Goubert L, Leinonen V. Protocol of identical exercise programs with and without specific breathing techniques for the treatment of chronic non-specific low back pain: randomized feasibility trial with two-month follow-up. BMC Musculoskelet Disord. 2023 May 5;24(1):354. doi: 10.1186/s12891-023-06434-6. PMID 37147638
- See also: Study web page — http://selkakuntoutus.fi/tutkimus-2022/